CLINICAL TRIAL: NCT00408408
Title: A Randomized Phase III Trial of Neoadjuvant Therapy in Patients With Palpable and Operable Breast Cancer Evaluating the Effect on Pathologic Complete Response (pCR) of Adding Capecitabine or Gemcitabine to Docetaxel When Administered Before AC With or Without Bevacizumab and Correlative Science Studies Attempting to Identify Predictors of High Likelihood for pCR With Each of the Regimens
Brief Title: Chemotherapy With or Without Bevacizumab in Treating Women With Stage I, Stage II, or Stage IIIA Breast Cancer That Can Be Removed By Surgery
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: NSABP Foundation Inc (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NSABP B-40; NSABP B-40
Record Dates: First submitted 2006-12-06; First posted 2006-12-07 (Estimated); Results first posted 2017-09-18 (Actual); Last update posted 2017-09-18 (Actual); Status verified 2017-09

CONDITIONS: Breast Cancer
Keywords: stage I breast cancer; stage II breast cancer; stage IIIA breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Bevacizumab; Capecitabine; Cyclophosphamide; Docetaxel; Doxorubicin; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Arm 1A: Docetaxel then AC (Active Comparator): Patients receive docetaxel IV on day 1 every 3 weeks for up to 4 cycles. Patients then receive AC IV every 3 weeks for up to 4 cycles. Patients then undergo surgery (lumpectomy or mastectomy).
  Interventions: Drug: cyclophosphamide; Drug: docetaxel; Drug: doxorubicin hydrochloride (Adriamycin)
- Arm 1B Docetaxel + Bev then AC + Bev (Experimental): Patients receive bevacizumab (bev) IV on day 1 and docetaxel every 3 weeks for up to 4 cycles. Patients then receive AC every 3 weeks for up to 4 cycles and 2 additional cycles of bevacizumab concurrent with the first 2 cycles of AC. Patients then undergo surgery as in Arm 1A. At least 4-6 weeks after surgery, patients receive adjuvant bevacizumab IV every 3 weeks for up to 10 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: bevacizumab; Drug: cyclophosphamide; Drug: docetaxel; Drug: doxorubicin hydrochloride (Adriamycin)
- Arm 2A: Docetaxel + Capecitabine then AC (Experimental): Patients receive docetaxel as in Arm 1A and oral capecitabine (cape) twice daily on days 1-14 every 3 weeks for up to 4 cycles. Patients then receive AC as in Arm 1A. Patients then undergo surgery as in Arm 1A.
  Interventions: Drug: capecitabine; Drug: cyclophosphamide; Drug: docetaxel; Drug: doxorubicin hydrochloride (Adriamycin)
- Arm 2B: Docetaxel + Cape + Bev then AC + Bev (Experimental): Patients receive bevacizumab as in Arm 1B and docetaxel and capecitabine as in Arm III. Treatment repeats every 3 weeks for up to 4 cycles. Patients then receive AC every 3 weeks for up to 4 cycles and 2 additional cycles of bevacizumab concurrent with the first 2 cycles of AC. Patients then undergo surgery as in Arm 1B. At least 4-6 weeks after surgery, patients receive adjuvant bevacizumab as in Arm 1B.
  Interventions: Biological: bevacizumab; Drug: capecitabine; Drug: cyclophosphamide; Drug: docetaxel; Drug: doxorubicin hydrochloride (Adriamycin)
- Arm 3A: Docetaxel + Gem then AC (Experimental): Patients receive docetaxel as in Arm 1A and gemcitabine hydrochloride IV on days 1 and 8 of each cycle every 3 weeks for up to 4 cycles. Patients then receive AC as in Arm 1A. Patients then undergo surgery as in Arm 1A.
  Interventions: Drug: cyclophosphamide; Drug: docetaxel; Drug: doxorubicin hydrochloride (Adriamycin); Drug: gemcitabine hydrochloride
- Arm 3B: Docetaxel + Gem + Bev then AC + Bev (Experimental): Patients receive docetaxel as in Arm 1A, gemcitabine hydrochloride as in Arm 3A, and bevacizumab as in Arm 1B. Patients then receive AC every 3 weeks for up to 4 cycles and 2 additional cycles of bevacizumab concurrent with the first 2 cycles of AC. Patients then undergo surgery as in Arm 1A. At least 4-6 weeks after surgery, patients receive adjuvant bevacizumab as in Arm 1B.
  Interventions: Biological: bevacizumab; Drug: cyclophosphamide; Drug: docetaxel; Drug: doxorubicin hydrochloride (Adriamycin); Drug: gemcitabine hydrochloride

INTERVENTIONS:
Biological: bevacizumab — 15 mg/kg IV
  Arms: Arm 1B Docetaxel + Bev then AC + Bev; Arm 2B: Docetaxel + Cape + Bev then AC + Bev; Arm 3B: Docetaxel + Gem + Bev then AC + Bev
Drug: capecitabine — 825 mg/m2 orally
  Arms: Arm 2A: Docetaxel + Capecitabine then AC; Arm 2B: Docetaxel + Cape + Bev then AC + Bev
Drug: cyclophosphamide — 600 mg/m2 IV
Drug: docetaxel — 100 mg/m2 IV
Drug: doxorubicin hydrochloride (Adriamycin) — 60 mg/m2 IV
Drug: gemcitabine hydrochloride — 1000 mg/m2 IV
  Arms: Arm 3A: Docetaxel + Gem then AC; Arm 3B: Docetaxel + Gem + Bev then AC + Bev

SUMMARY:
RATIONALE: Drugs used in chemotherapy work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more tumor cells. Monoclonal antibodies, such as bevacizumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Bevacizumab may also stop the growth of breast cancer by blocking blood flow to the tumor. Giving chemotherapy and bevacizumab before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed. Giving bevacizumab after surgery may kill any tumor cells that remain after surgery. It is not yet known which chemotherapy regimen is more effective with or without bevacizumab in treating breast cancer.

PURPOSE: This randomized phase III trial is studying six different chemotherapy regimens to compare how well they work with or without bevacizumab in treating women with stage I, stage II, or stage IIIA breast cancer that can be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the efficacy of docetaxel followed by doxorubicin hydrocloride and cyclophosphamide (AC) vs docetaxel and capecitabine followed by AC vs docetaxel and gemcitabine hydrochloride followed by AC, with or without bevacizumab, in terms of an increase in the rate of pathologic complete response (pCR) in the breast, in women with palpable or operable breast cancer.

Secondary

* Compare docetaxel/capecitabine with AC vs docetaxel/gemcitabine hydrochloride with AC vs docetaxel with AC, with or without bevacizumab, in terms of the rate of pCR in the breast and all post-therapy lymph nodes evaluated histologically (pCR breast and nodes).
* Determine whether the addition of bevacizumab to the docetaxel/anthracycline-based regimens (docetaxel with AC, docetaxel and capecitabine with AC, and docetaxel and gemcitabine hydrochloride with AC) will increase the rate of pCR of the breast and nodes compared to the same docetaxel/anthracycline-based regimens without bevacizumab in these patients.
* Determine whether the addition of capecitabine or gemcitabine hydrochloride to docetaxel, with or without bevacizumab, will increase the rate of clinical overall response (cOR) compared to docetaxel alone with or without bevacizumab in these patients.
* Determine whether the addition of bevacizumab to the docetaxel/anthracycline-based regimens will increase the rate of cOR compared to the same docetaxel/anthracycline-based regimens without bevacizumab in these patients.
* Determine whether the addition of capecitabine or gemcitabine hydrochloride to docetaxel, with or without bevacizumab, will increase the rate of clinical complete response (cCR) compared to docetaxel alone with or without bevacizumab in these patients.
* Determine whether the addition of bevacizumab to the docetaxel/anthracycline-based regimens (docetaxel with AC, docetaxel/capecitabine with AC, and docetaxel/gemcitabine hydrochloride with AC) will increase the rate of cCR compared to the same docetaxel/anthracycline-based regimens without bevacizumab in these patients.
* Identify gene expression profiles that can predict pCR in patients treated with the different sequential docetaxel/anthracycline-based regimens with or without bevacizumab.
* Identify gene expression profiles that can predict cOR in patients treated with docetaxel alone, docetaxel/capecitabine, or docetaxel/gemcitabine hydrochloride with or without bevacizumab.
* Determine the accuracy of an in vitro chemoresponse assay (ChemoFx®) as a predictor of pCR in patients treated with the different sequential docetaxel/anthracycline-based regimens without bevacizumab.
* Determine the accuracy of ChemoFx® as a predictor of cOR in patients treated with docetaxel alone, docetaxel/capecitabine, or docetaxel/gemcitabine hydrochloride without bevacizumab in these patients.
* Determine the impact of preoperative bevacizumab and sequential chemotherapy regimens and postoperative bevacizumab therapy on cardiac function in these patients.
* Determine the impact of bevacizumab on surgical complications in these patients.
* Determine the toxicity of the preoperative regimens and the toxicity of postoperative bevacizumab in these patients.
* Compare the docetaxel/anthracycline-based regimens with vs without bevacizumab, in terms of an increase in disease-free survival, of these patients.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to tumor size (2-4 cm vs > 4 cm), nodal status (negative vs positive), hormone receptor status (estrogen receptor [ER]-positive and/or progesterone-receptor [PgR]-positive vs ER- and PgR-negative), and age (< 50 years vs ≥ 50 years). Patients are randomized to 1 of 6 treatment arms.

Core needle biopsies are performed at baseline. Tumor tissue samples are also collected during definitive surgery. Samples are examined for gene expression and polymorphism by reverse transcriptase-polymerase chain reaction analysis and chemoresponse assay (ChemoFx®).

After completion of study therapy, patients are followed periodically for 10 years.

PROJECTED ACCRUAL: A total of 1,200 patients will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria:

* The patient must have consented to participate and must have signed and dated an appropriate Institutional Review Board (IRB)-approved consent form that conforms to federal and institutional guidelines for the study treatment and submission of pre-entry core biopsy material for correlative studies.
* Patients must be female.
* Patients must be 18 years of age or older.
* Patients must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* The diagnosis of invasive adenocarcinoma of the breast must have been made by core needle biopsy.
* The primary breast tumor must be palpable and measure greater than or equal to 2.0 cm on physical exam.
* All patients must have their left ventricular ejection fraction (LVEF) assessed by multigated acquisition (MUGA) scan or echocardiogram within 3 months prior to study entry. The LVEF must be greater than or equal to the lower limit of normal (LLN) for the cardiac imaging facility performing the study. Note: If the cardiac imaging facility cannot provide a LLN, use 50% as the LLN value.

  - Note: Since the pre-entry LVEF serves as the baseline for comparing subsequent LVEF assessments to determine if bevacizumab therapy can be continued, it is critical that this baseline study be an accurate assessment of the patient's LVEF. If the baseline LVEF is greater than 75%, the investigator should have the study reviewed for accuracy prior to study entry. Following study entry, the LVEF determination may be reviewed up until the time of the post-chemotherapy (preoperative) evaluation. Please note that if a more accurate value is obtained from the review of the baseline MUGA or echocardiogram, the correct value must be submitted to the NSABP before the post-chemotherapy (preoperative) MUGA or echocardiogram is performed or it cannot be used for managing postoperative bevacizumab.
* All patients must have an EKG within 3 months prior to study entry.
* At the time of randomization:

  * Absolute neutrophil count (ANC) must be greater than or equal to 1200/mm3.
  * Platelet count must be greater than or equal to 100,000/mm3.
  * Hemoglobin must be greater than or equal to 10 g/dL.
  * There must be evidence of adequate hepatic function by these criteria:
  * Total bilirubin must be less than or equal to the ULN for the lab unless the patient has a grade 1 bilirubin elevation (greater than ULN to 1.5 x ULN) resulting from Gilbert's disease or similar syndrome due to slow conjugation of bilirubin; and
  * Alkaline phosphatase must be less than or equal 2.5 x ULN for the lab; and
  * Aspartate Aminotransferase (AST) must be less than or equal to 1.5 x ULN for the lab.
  * Alkaline phosphatase and AST may not both be greater than the ULN. For example, if the alkaline phosphatase is greater than the ULN but less than or equal 2.5 x ULN, then the AST must be less than or equal the ULN. If the AST is greater than the ULN but less than or equal 1.5 x ULN, then the alkaline phosphatase must be less than or equal ULN.
* Patients with either skeletal pain or alkaline phosphatase that is greater than ULN but less than or equal 2.5 x ULN are eligible for inclusion in the study if bone scans do not demonstrate metastatic disease. Suspicious findings on bone scan must be confirmed as benign by x-ray, MRI, or biopsy.
* Patients with AST or alkaline phosphatase greater than ULN are eligible for inclusion in the study if liver imaging does not demonstrate metastatic disease and adequate bone marrow and liver function results as described above are met.
* The following criteria for evidence of adequate renal function must be met:
* Serum creatinine less than or equal ULN for the lab.
* Calculated creatinine clearance must be greater than 50 mL/min.
* Urine protein/urine creatinine (UPC) ratio must be less than 1.0.
* Patient must be able to swallow oral medications.

Exclusion criteria:

* Tumor determined to be strongly human epidermal growth factor receptor 2 (HER2)-positive by immunohistochemistry (3+) or by fluorescent in situ hybridization (positive for gene amplification).
* Excisional or incisional biopsy for this primary breast tumor.
* Surgical axillary staging procedure prior to study entry. Exceptions: 1) Fine Needle Aspiration (FNA) or core biopsy of an axillary node is permitted for any patient, and 2) although not recommended, a pre-neoadjuvant therapy sentinel lymph node biopsy for patients with clinically negative axillary nodes is permitted.
* Tumors clinically staged as T4.
* Ipsilateral cN2b or cN3 disease. (Patients with cN1 or cN2a disease are eligible.)
* Definitive clinical or radiologic evidence of metastatic disease.
* Synchronous bilateral breast cancer (invasive or DCIS).
* Treatment including radiation therapy, chemotherapy, biotherapy, and/or hormonal therapy for the currently diagnosed breast cancer prior to study entry.
* Any sex hormonal therapy, e.g., birth control pills, ovarian hormonal replacement therapy, etc. (These patients are eligible if this therapy is discontinued prior to randomization.)
* Therapy with any hormonal agent such as raloxifene, tamoxifen, or other selective estrogen receptor modulator (SERM), either for osteoporosis or breast cancer prevention. (Patients are eligible only if these medications are discontinued prior to randomization.)
* Prior history of breast cancer, including DCIS. (Patients with a history of lobular carcinoma in situ [LCIS] are eligible.)
* Prior therapy with anthracyclines, taxanes, capecitabine, 5-FU (fluorouracil), gemcitabine, or bevacizumab for any malignancy.
* Other malignancies unless the patient is considered to be disease-free for 5 or more years prior to randomization and is deemed by her physician to be at low risk for recurrence. Patients with the following cancers are eligible if diagnosed and treated within the past 5 years: carcinoma in situ of the cervix, carcinoma in situ of the colon, melanoma in situ, and basal cell and squamous cell carcinoma of the skin.
* Cardiac disease that would preclude the use of anthracyclines. This includes:

  * angina pectoris that requires the use of anti-anginal medication;
  * history of documented congestive heart failure;
  * serious cardiac arrhythmia requiring medication;
  * severe conduction abnormality;
  * valvular disease with documented cardiac function compromise; and
  * uncontrolled hypertension defined as BP greater than 150/90 on antihypertensive therapy. (Patients with hypertension that is well controlled on medication are eligible.)
* History of myocardial infarction documented by elevated cardiac enzymes or persistent regional wall abnormalities on assessment of LV function.
* History of transient ischemic attack (TIA) or cerebrovascular accident (CVA).
* History of other arterial thrombotic event within 12 months before study entry.
* Symptomatic peripheral vascular disease.
* Any significant non-traumatic bleeding within 6 months before study entry.
* Serious or non-healing wound, skin ulcers, or incompletely healed bone fracture.
* Gastroduodenal ulcer(s) determined by endoscopy to be active.
* Invasive procedures defined as follows:

  * Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to planned start of study therapy. (Note: Placement of a vascular access device is not considered a major surgical procedure.)
  * Anticipation of need for major surgical procedures (other than the required breast surgery) during the course of the study.
* Known bleeding diathesis or coagulopathy. (Patients on warfarin with an in-range international normalized ratio [INR] [usually between 2 and 3] are eligible.)
* Sensory/motor neuropathy greater than or equal grade 2, as defined by the NCI's Common Terminology Criteria for Adverse Events Version 3.0 (CTCAE v3.0).
* Other non-malignant systemic disease (cardiovascular, renal, hepatic, etc.) that would preclude treatment with any of the treatment regimens or would prevent required follow-up.
* Conditions that would prohibit administration of corticosteroids.
* History of severe hypersensitivity reaction to drugs formulated with polysorbate 80.
* Administration of any investigational agents within 30 days before study entry.
* Pregnancy or lactation at the time of proposed randomization.

Ages: 18 Years to 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1206 (Actual)
Dates: Start 2006-11; Primary Completion 2011-03 (Actual); Study Completion 2018-03 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Norman Wolmark, MD, Principal Investigator — NSABP Foundation Inc
Locations (442):
- United States (432):
  - Arkansas Cancer Research Center at University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - East Bay Radiation Oncology Center, Castro Valley, California
  - Eden Medical Center, Castro Valley, California
  - Valley Medical Oncology Consultants - Castro Valley, Castro Valley, California
  - Kaiser Permanente - Fremont, Fremont, California
  - Valley Medical Oncology, Fremont, California
  - Cancer Care Associates, Fresno, California
  - Kaiser Permanente Medical Center - Hayward, Hayward, California
  - Scripps Cancer Center - San Diego, La Jolla, California
  - Loma Linda University Cancer Institute at Loma Linda University Medical Center, Loma Linda, California
  - Contra Costa Regional Medical Center, Martinez, California
  - El Camino Hospital Cancer Center, Mountain View, California
  - Highland General Hospital, Oakland, California
  - Alta Bates Summit Medical Center - Summit Campus, Oakland, California
  - Bay Area Breast Surgeons, Incorporated, Oakland, California
  - CCOP - Bay Area Tumor Institute, Oakland, California
  - Larry G Strieff MD Medical Corporation, Oakland, California
  - Tom K Lee, Incorporated, Oakland, California
  - Kaiser Permanente Medical Center - Oakland, Oakland, California
  - St. Joseph Hospital Regional Cancer Center - Orange, Orange, California
  - Desert Regional Medical Center Comprehensive Cancer Center, Palm Springs, California
  - Valley Care Medical Center, Pleasanton, California
  - Valley Medical Oncology Consultants - Pleasanton, Pleasanton, California
  - Kaiser Permanente Medical Center - Redwood City, Redwood City, California
  - Kaiser Permanente Medical Center - Richmond, Richmond, California
  - Kaiser Permanente Medical Center - Roseville, Roseville, California
  - South Sacramento Kaiser-Permanente Medical Center, Sacramento, California
  - Kaiser Permanente Medical Center - Sacramento, Sacramento, California
  - Salinas Valley Memorial Hospital, Salinas, California
  - Kaiser Permanente Medical Office -Vandever Medical Office, San Diego, California
  - Kaiser Permanente Medical Center - San Francisco Geary Campus, San Francisco, California
  - Kaiser Permanente Medical Center - Santa Teresa, San Jose, California
  - Doctors Medical Center - San Pablo Campus, San Pablo, California
  - Kaiser Foundation Hospital - San Rafael, San Rafael, California
  - Kaiser Permanente Medical Center - Santa Clara Kiely Campus, Santa Clara, California
  - Kaiser Permanente Medical Center - Santa Rosa, Santa Rosa, California
  - Kaiser Permanente Medical Center - South San Francisco, South San Francisco, California
  - Kaiser Permanente Medical Facility - Stockton, Stockton, California
  - Kaiser Permanente Medical Center - Vallejo, Vallejo, California
  - Kaiser Permanente Medical Center - Walnut Creek, Walnut Creek, California
  - Aurora Presbyterian Hospital, Aurora, Colorado
  - Boulder Community Hospital, Boulder, Colorado
  - Memorial Hospital Cancer Center - Colorado Springs, Colorado Springs, Colorado
  - Penrose Cancer Center at Penrose Hospital, Colorado Springs, Colorado
  - St. Anthony Central Hospital, Denver, Colorado
  - Kaiser Permanente - Denver, Denver, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Presbyterian - St. Luke's Medical Center, Denver, Colorado
  - St. Joseph Hospital, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - CCOP - Colorado Cancer Research Program, Denver, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - St. Mary's Regional Cancer Center at St. Mary's Hospital and Medical Center, Grand Junction, Colorado
  - North Colorado Medical Center, Greeley, Colorado
  - Kaiser Permanente - Lafayette, Lafayette, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Hope Cancer Care Center at Longmont United Hospital, Longmont, Colorado
  - McKee Medical Center, Loveland, Colorado
  - St. Mary - Corwin Regional Medical Center, Pueblo, Colorado
  - North Suburban Medical Center, Thornton, Colorado
  - Exempla Lutheran Medical Center, Wheat Ridge, Colorado
  - Carole and Ray Neag Comprehensive Cancer Center at the University of Connecticut Health Center, Farmington, Connecticut
  - Helen and Harry Gray Cancer Center at Hartford Hospital, Hartford, Connecticut
  - Saint Francis/Mount Sinai Regional Cancer Center at Saint Francis Hospital and Medical Center, Hartford, Connecticut
  - Eastern Connecticut Hematology and Oncology Associates, Norwich, Connecticut
  - Tunnell Cancer Center at Beebe Medical Center, Lewes, Delaware
  - CCOP - Christiana Care Health Services, Newark, Delaware
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - Herbert D. Kerman Regional Oncology Center - Daytona Beach, Daytona Beach, Florida
  - Michael and Dianne Bienes Comprehensive Cancer Center at Holy Cross Hospital, Fort Lauderdale, Florida
  - Broward General Medical Center Cancer Center, Fort Lauderdale, Florida
  - Baptist Cancer Institute - Jacksonville, Jacksonville, Florida
  - Ella Milbank Foshay Cancer Center at Jupiter Medical Center, Jupiter, Florida
  - CCOP - Mount Sinai Medical Center, Miami Beach, Florida
  - Florida Hospital Cancer Institute at Florida Hospital Orlando, Orlando, Florida
  - M.D. Anderson Cancer Center at Orlando, Orlando, Florida
  - Phoebe Cancer Center at Phoebe Putney Memorial Hospital, Albany, Georgia
  - Northeast Georgia Medical Center, Gainesville, Georgia
  - Curtis and Elizabeth Anderson Cancer Institute at Memorial Health University Medical Center, Savannah, Georgia
  - Nancy N. and J. C. Lewis Cancer and Research Pavilion at St. Joseph's/Candler, Savannah, Georgia
  - Cancer Research Center of Hawaii, Honolulu, Hawaii
  - OnCare Hawaii, Incorporated - Lusitana, Honolulu, Hawaii
  - Queen's Cancer Institute at Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Incorporated, Honolulu, Hawaii
  - Hawaii Medical Center - East, Honolulu, Hawaii
  - OnCare Hawaii, Incorporated - Kuakini, Honolulu, Hawaii
  - Kaiser Permanente - Moanalua Medical Center and Clinic, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Maui Memorial Medical Center, Wailuku, Hawaii
  - Pacific Cancer Institute - Maui, Wailuku, Hawaii
  - Kapiolani Medical Center at Pali Momi, ‘Aiea, Hawaii
  - Kootenai Cancer Center - Coeur d'Alene, Coeur d'Alene, Idaho
  - Saint Anthony's Hospital at Saint Anthony's Health Center, Alton, Illinois
  - Illinois CancerCare - Bloomington, Bloomington, Illinois
  - St. Joseph Medical Center, Bloomington, Illinois
  - Graham Hospital, Canton, Illinois
  - Illinois CancerCare - Canton, Canton, Illinois
  - Illinois CancerCare - Carthage, Carthage, Illinois
  - Memorial Hospital, Carthage, Illinois
  - Mount Sinai Hospital Medical Center, Chicago, Illinois
  - John H. Stroger, Jr. Hospital of Cook County, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - Decatur Memorial Hospital Cancer Care Institute, Decatur, Illinois
  - Alexian Brothers Radiation Oncology, Elk Grove Village, Illinois
  - Eureka Community Hospital, Eureka, Illinois
  - Illinois CancerCare - Eureka, Eureka, Illinois
  - St. Francis Hospital, Evanston, Illinois
  - Galesburg Clinic, PC, Galesburg, Illinois
  - Galesburg Cottage Hospital, Galesburg, Illinois
  - Illinois CancerCare - Cottage, Galesburg, Illinois
  - Illinois CancerCare - Galesburg, Galesburg, Illinois
  - Illinois CancerCare - Havana, Havana, Illinois
  - Mason District Hospital, Havana, Illinois
  - Illinois CancerCare - Kewanee Clinic, Kewanee, Illinois
  - Illinois CancerCare - Macomb, Macomb, Illinois
  - McDonough District Hospital, Macomb, Illinois
  - Cardinal Bernardin Cancer Center at Loyola University Medical Center, Maywood, Illinois
  - Illinois CancerCare - Monmouth, Monmouth, Illinois
  - OSF Holy Family Medical Center, Monmouth, Illinois
  - Good Samaritan Regional Health Center, Mount Vernon, Illinois
  - Edward Hospital Cancer Center, Naperville, Illinois
  - BroMenn Regional Medical Center, Normal, Illinois
  - Community Cancer Center, Normal, Illinois
  - Illinois CancerCare - Community Cancer Center, Normal, Illinois
  - Community Hospital of Ottawa, Ottawa, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Ottawa, Ottawa, Illinois
  - Illinois CancerCare - Pekin, Pekin, Illinois
  - Proctor Hospital, Peoria, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF St. Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare - Peru, Peru, Illinois
  - Illinois Valley Community Hospital, Peru, Illinois
  - Illinois CancerCare - Princeton, Princeton, Illinois
  - Perry Memorial Hospital, Princeton, Illinois
  - Swedish-American Regional Cancer Center, Rockford, Illinois
  - Illinois CancerCare - Spring Valley, Spring Valley, Illinois
  - Regional Cancer Center at Memorial Medical Center, Springfield, Illinois
  - St. Francis Hospital and Health Centers - Beech Grove Campus, Beech Grove, Indiana
  - Elkhart Clinic, LLC, Elkhart, Indiana
  - Elkhart General Hospital, Elkhart, Indiana
  - Fort Wayne Medical Oncology and Hematology, Fort Wayne, Indiana
  - Center for Cancer Care at Goshen General Hospital, Goshen, Indiana
  - St. Vincent Indianapolis Hospital, Indianapolis, Indiana
  - Howard Community Hospital, Kokomo, Indiana
  - Center for Cancer Therapy at LaPorte Hospital and Health Services, La Porte, Indiana
  - Community Hospital, Munster, Indiana
  - Reid Hospital & Health Care Services, Richmond, Indiana
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Michiana Hematology-Oncology, PC - South Bend, South Bend, Indiana
  - Saint Joseph Regional Medical Center, South Bend, Indiana
  - South Bend Clinic, South Bend, Indiana
  - McFarland Clinic, PC, Ames, Iowa
  - Holden Comprehensive Cancer Center at University of Iowa, Iowa City, Iowa
  - Cancer Center of Kansas, PA - Chanute, Chanute, Kansas
  - Cancer Center of Kansas, PA - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas, PA - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Cancer Center of Kansas, PA - Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Southwest Medical Center, Liberal, Kansas
  - Cancer Center of Kansas, PA - Newton, Newton, Kansas
  - Menorah Medical Center, Overland Park, Kansas
  - Saint Luke's Hospital - South, Overland Park, Kansas
  - Cancer Center of Kansas, PA - Parsons, Parsons, Kansas
  - Cancer Center of Kansas, PA - Pratt, Pratt, Kansas
  - Cancer Center of Kansas, PA - Salina, Salina, Kansas
  - Shawnee Mission Medical Center, Shawnee, Kansas
  - Cancer Center of Kansas, PA - Wellington, Wellington, Kansas
  - Associates in Womens Health, PA - North Review, Wichita, Kansas
  - Cancer Center of Kansas, PA - Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas, PA - Wichita, Wichita, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Cancer Center at Via Christi Regional Medical Center, Wichita, Kansas
  - Wesley Medical Center, Wichita, Kansas
  - Cancer Center of Kansas, PA - Winfield, Winfield, Kansas
  - Cancer Resource Center at King's Daughters Medical Center, Ashland, Kentucky
  - Lucille P. Markey Cancer Center at University of Kentucky, Lexington, Kentucky
  - Louisville Oncology at Norton Cancer Institute - Louisville, Louisville, Kentucky
  - James Graham Brown Cancer Center at University of Louisville, Louisville, Kentucky
  - Mary Bird Perkins Cancer Center - Baton Rouge, Baton Rouge, Louisiana
  - Ochsner Health Center - Bluebonnet, Baton Rouge, Louisiana
  - MBCCOP - LSU Health Sciences Center, New Orleans, Louisiana
  - Medical Center of Louisiana - New Orleans, New Orleans, Louisiana
  - CCOP - Ochsner, New Orleans, Louisiana
  - Ochsner Cancer Institute at Ochsner Clinic Foundation, New Orleans, Louisiana
  - York Hospital's Oncology Treatment Center, York Village, Maine
  - Greenebaum Cancer Center at University of Maryland Medical Center, Baltimore, Maryland
  - Greater Baltimore Medical Center Cancer Center, Baltimore, Maryland
  - St. Agnes Hospital Cancer Center, Baltimore, Maryland
  - Harry & Jeanette Weinberg Cancer Institute at Franklin Square Hospital Center, Baltimore, Maryland
  - Frederick Memorial Hospital Regional Cancer Therapy Center, Frederick, Maryland
  - Associates in Oncology and Hematology - Medical Center Drive, Rockville, Maryland
  - Peninsula Regional Medical Center, Salisbury, Maryland
  - MetroWest Medical Center - Framingham Union Hospital, Framingham, Massachusetts
  - Hickman Cancer Center at Bixby Medical Center, Adrian, Michigan
  - Saint Joseph Mercy Cancer Center, Ann Arbor, Michigan
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - Oakwood Cancer Center at Oakwood Hospital and Medical Center, Dearborn, Michigan
  - Josephine Ford Cancer Center at Henry Ford Hospital, Detroit, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Great Lakes Cancer Institute at McLaren Regional Medical Center, Flint, Michigan
  - Van Elslander Cancer Center at St. John Hospital and Medical Center, Grosse Pointe Woods, Michigan
  - Foote Memorial Hospital, Jackson, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Haematology-Oncology Associates of Ohio and Michigan, PC, Lambertville, Michigan
  - Breslin Cancer Center at Ingham Regional Medical Center, Lansing, Michigan
  - Sparrow Regional Cancer Center, Lansing, Michigan
  - Lapeer Regional Hospital, Lapeer, Michigan
  - St. Mary Mercy Hospital, Livonia, Michigan
  - Community Cancer Center of Monroe, Monroe, Michigan
  - Mercy Memorial Hospital - Monroe, Monroe, Michigan
  - St. Joseph Mercy Oakland, Pontiac, Michigan
  - Mercy Regional Cancer Center at Mercy Hospital, Port Huron, Michigan
  - Seton Cancer Institute at Saint Mary's - Saginaw, Saginaw, Michigan
  - Lakeland Regional Cancer Care Center - St. Joseph, Saint Joseph, Michigan
  - Lakeside Cancer Specialists, PLLC, Saint Joseph, Michigan
  - Providence Cancer Institute at Providence Hospital - Southfield Campus, Southfield, Michigan
  - St. John Macomb Hospital, Warren, Michigan
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy and Unity Cancer Center at Mercy Hospital, Coon Rapids, Minnesota
  - Duluth Clinic Cancer Center - Duluth, Duluth, Minnesota
  - CCOP - Duluth, Duluth, Minnesota
  - Miller - Dwan Medical Center, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Mercy and Unity Cancer Center at Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - HealthEast Cancer Care at St. John's Hospital, Maplewood, Minnesota
  - Minnesota Oncology Hematology, PA - Maplewood, Maplewood, Minnesota
  - Virginia Piper Cancer Institute at Abbott - Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center - Minneapolis, Minneapolis, Minnesota
  - Hubert H. Humphrey Cancer Center at North Memorial Outpatient Center, Robbinsdale, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Park Nicollet Cancer Center, Saint Louis Park, Minnesota
  - Regions Hospital Cancer Care Center, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - St. Francis Cancer Center at St. Francis Medical Center, Shakopee, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Minnesota Oncology Hematology, PA - Woodbury, Woodbury, Minnesota
  - Hattiesburg Clinic, PA at Forrest General, Hattiesburg, Mississippi
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Ellis Fischel Cancer Center at University of Missouri - Columbia, Columbia, Missouri
  - St. John's Regional Medical Center, Joplin, Missouri
  - Truman Medical Center - Hospital Hill, Kansas City, Missouri
  - Saint Luke's Cancer Institute at Saint Luke's Hospital, Kansas City, Missouri
  - St. Joseph Medical Center, Kansas City, Missouri
  - North Kansas City Hospital, Kansas City, Missouri
  - Parvin Radiation Oncology, Kansas City, Missouri
  - Heartland Hematology Oncology Associates, Incorporated, Kansas City, Missouri
  - CCOP - Kansas City, Kansas City, Missouri
  - Research Medical Center, Kansas City, Missouri
  - Saint Luke's East - Lee's Summit, Lee's Summit, Missouri
  - Liberty Hospital, Liberty, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - St. John's Regional Health Center, Springfield, Missouri
  - Hulston Cancer Center at Cox Medical Center South, Springfield, Missouri
  - Midwest Hematology Oncology Group, Incorporated, St Louis, Missouri
  - Saint Louis University Cancer Center, St Louis, Missouri
  - CCOP - St. Louis-Cape Girardeau, St Louis, Missouri
  - David C. Pratt Cancer Center at St. John's Mercy, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Hematology-Oncology Centers of the Northern Rockies - Billings, Billings, Montana
  - Northern Rockies Radiation Oncology Center, Billings, Montana
  - St. Vincent Healthcare Cancer Care Services, Billings, Montana
  - Billings Clinic - Downtown, Billings, Montana
  - Bozeman Deaconess Cancer Center, Bozeman, Montana
  - St. James Healthcare Cancer Care, Butte, Montana
  - Big Sky Oncology, Great Falls, Montana
  - Great Falls Clinic - Main Facility, Great Falls, Montana
  - Sletten Cancer Institute at Benefis Healthcare, Great Falls, Montana
  - Great Falls, Montana
  - St. Peter's Hospital, Helena, Montana
  - Glacier Oncology, PLLC, Kalispell, Montana
  - Kalispell Medical Oncology at KRMC, Kalispell, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Community Medical Center, Missoula, Montana
  - Guardian Oncology and Center for Wellness, Missoula, Montana
  - Montana Cancer Specialists at Montana Cancer Center, Missoula, Montana
  - Montana Cancer Center at St. Patrick Hospital and Health Sciences Center, Missoula, Montana
  - Good Samaritan Cancer Center at Good Samaritan Hospital, Kearney, Nebraska
  - Cancer Resource Center - Lincoln, Lincoln, Nebraska
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Immanuel Medical Center, Omaha, Nebraska
  - Alegant Health Cancer Center at Bergan Mercy Medical Center, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - Cancer Institute of New Jersey at Hamilton, Hamilton, New Jersey
  - Cancer Institute of New Jersey at UMDNJ - Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Cancer Institute of New Jersey at Cooper - Voorhees, Voorhees Township, New Jersey
  - Charles R. Wood Cancer Center at Glens Falls Hospital, Glens Falls, New York
  - Tucker Center for Cancer Care at Orange Regional Medical Center, Middletown, New York
  - Saint Francis Hospital Cancer Center, Poughkeepsie, New York
  - Our Lady of Mercy Medical Center Comprehensive Cancer Center, The Bronx, New York
  - Randolph Hospital, Asheboro, North Carolina
  - Hope A Women's Cancer Center, Asheville, North Carolina
  - Alamance Cancer Center at Alamance Regional Medical Center, Burlington, North Carolina
  - Blumenthal Cancer Center at Carolinas Medical Center, Charlotte, North Carolina
  - Presbyterian Cancer Center at Presbyterian Hospital, Charlotte, North Carolina
  - Batte Cancer Center at Northeast Medical Center, Concord, North Carolina
  - Wayne Memorial Hospital, Incorporated, Goldsboro, North Carolina
  - Moses Cone Regional Cancer Center at Wesley Long Community Hospital, Greensboro, North Carolina
  - Annie Penn Cancer Center, Reidsville, North Carolina
  - Rutherford Hospital, Rutherfordton, North Carolina
  - Iredell Memorial Hospital, Statesville, North Carolina
  - Marion L. Shepard Cancer Center at Beaufort County Hospital, Washington, North Carolina
  - Forsyth Regional Cancer Center at Forsyth Medical Center, Winston-Salem, North Carolina
  - Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina
  - Altru Cancer Center at Altru Hospital, Grand Forks, North Dakota
  - McDowell Cancer Center at Akron General Medical Center, Akron, Ohio
  - Summa Center for Cancer Care at Akron City Hospital, Akron, Ohio
  - Barberton Citizens Hospital, Barberton, Ohio
  - Wood County Oncology Center, Bowling Green, Ohio
  - Aultman Cancer Center at Aultman Hospital, Canton, Ohio
  - Case Comprehensive Cancer Center, Cleveland, Ohio
  - North Coast Cancer Care - Clyde, Clyde, Ohio
  - Arthur G. James Cancer Hospital and Richard J. Solove Research Institute at Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital, Dayton, Ohio
  - David L. Rike Cancer Center at Miami Valley Hospital, Dayton, Ohio
  - Samaritan North Cancer Care Center, Dayton, Ohio
  - CCOP - Dayton, Dayton, Ohio
  - Community Cancer Center, Elyria, Ohio
  - Hematology Oncology Center, Elyria, Ohio
  - Blanchard Valley Medical Associates, Findlay, Ohio
  - Middletown Regional Hospital, Franklin, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Charles F. Kettering Memorial Hospital, Kettering, Ohio
  - Lima Memorial Hospital, Lima, Ohio
  - Northwest Ohio Oncology Center, Maumee, Ohio
  - St. Luke's Hospital, Maumee, Ohio
  - Fisher-Titus Medical Center, Norwalk, Ohio
  - St. Charles Mercy Hospital, Oregon, Ohio
  - Toledo Clinic - Oregon, Oregon, Ohio
  - Cancer Care Center, Incorporated, Salem, Ohio
  - North Coast Cancer Care, Incorporated, Sandusky, Ohio
  - Flower Hospital Cancer Center, Sylvania, Ohio
  - Mercy Hospital of Tiffin, Tiffin, Ohio
  - Toledo Hospital, Toledo, Ohio
  - St. Vincent Mercy Medical Center, Toledo, Ohio
  - Medical University of Ohio Cancer Center, Toledo, Ohio
  - CCOP - Toledo Community Hospital, Toledo, Ohio
  - St. Anne Mercy Hospital, Toledo, Ohio
  - Toledo Clinic, Incorporated - Main Clinic, Toledo, Ohio
  - UVMC Cancer Care Center at Upper Valley Medical Center, Troy, Ohio
  - Fulton County Health Center, Wauseon, Ohio
  - Clinton Memorial Hospital, Wilmington, Ohio
  - Cancer Treatment Center, Wooster, Ohio
  - Ruth G. McMillan Cancer Center at Greene Memorial Hospital, Xenia, Ohio
  - Cleo Craig Cancer Research Clinic, Lawton, Oklahoma
  - Kaiser Permanente Health Care - Portland, Portland, Oregon
  - Morgan Cancer Center at Lehigh Valley Hospital - Cedar Crest, Allentown, Pennsylvania
  - St. Luke's Cancer Network at St. Luke's Hospital, Bethlehem, Pennsylvania
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Geisinger Cancer Institute at Geisinger Health, Danville, Pennsylvania
  - Cherry Tree Cancer Center, Hanover, Pennsylvania
  - Penn State Cancer Institute at Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Cancer Center of Paoli Memorial Hospital, Paoli, Pennsylvania
  - Allegheny Cancer Center at Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Western Pennsylvania Cancer Institute at Western Pennsylvania Hospital, Pittsburgh, Pennsylvania
  - UPMC Cancer Centers, Pittsburgh, Pennsylvania
  - McGlinn Family Regional Cancer Center at Reading Hospital and Medical Center, Reading, Pennsylvania
  - Geisinger Medical Group - Scenery Park, State College, Pennsylvania
  - Mount Nittany Medical Center, State College, Pennsylvania
  - Frank M. and Dorothea Henry Cancer Center at Geisinger Wyoming Valley Medical Center, Wilkes-Barre, Pennsylvania
  - CCOP - Main Line Health, Wynnewood, Pennsylvania
  - Lankenau Cancer Center at Lankenau Hospital, Wynnewood, Pennsylvania
  - York Cancer Center at Apple Hill Medical Center, York, Pennsylvania
  - AnMed Cancer Center, Anderson, South Carolina
  - Roper St. Francis Cancer Center at Roper Hospital, Charleston, South Carolina
  - Hollings Cancer Center at Medical University of South Carolina, Charleston, South Carolina
  - CCOP - Greenville, Greenville, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Gibbs Regional Cancer Center at Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - Medical X-Ray Center, PC, Sioux Falls, South Dakota
  - Sanford Cancer Center at Sanford USD Medical Center, Sioux Falls, South Dakota
  - Thompson Cancer Survival Center, Knoxville, Tennessee
  - University of Tennessee Cancer Institute - Memphis, Memphis, Tennessee
  - Nashville Oncology Associates, PC, Nashville, Tennessee
  - MBCCOP - Meharry Medical College - Nashville, Nashville, Tennessee
  - Doctor's Hospital of Laredo, Laredo, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - American Fork Hospital, American Fork, Utah
  - Sandra L. Maxwell Cancer Center, Cedar City, Utah
  - Jon and Karen Huntsman Cancer Center at Intermountain Medical Center, Murray, Utah
  - Val and Ann Browning Cancer Center at McKay-Dee Hospital Center, Ogden, Utah
  - Utah Valley Regional Medical Center - Provo, Provo, Utah
  - LDS Hospital, Salt Lake City, Utah
  - Utah Cancer Specialists at UCS Cancer Center, Salt Lake City, Utah
  - Huntsman Cancer Institute at University of Utah, Salt Lake City, Utah
  - Dixie Regional Medical Center - East Campus, St. George, Utah
  - Mountainview Medical, Berlin Corners, Vermont
  - Fletcher Allen Health Care - University Health Center Campus, Burlington, Vermont
  - Fredericksburg Oncology, Incorporated, Fredericksburg, Virginia
  - Virginia Commonwealth University Massey Cancer Center, Richmond, Virginia
  - Auburn Regional Center for Cancer Care, Auburn, Washington
  - Providence Centralia Hospital, Centralia, Washington
  - St. Francis Hospital, Federal Way, Washington
  - Providence St. Peter Hospital Regional Cancer Center, Olympia, Washington
  - Good Samaritan Cancer Center, Puyallup, Washington
  - Franciscan Cancer Center at St. Joseph Medical Center, Tacoma, Washington
  - Allenmore Hospital, Tacoma, Washington
  - CCOP - Northwest, Tacoma, Washington
  - MultiCare Regional Cancer Center at Tacoma General Hospital, Tacoma, Washington
  - St. Clare Hospital, Tacoma, Washington
  - West Virginia University Health Sciences Center - Charleston, Charleston, West Virginia
  - Mary Babb Randolph Cancer Center at West Virginia University Hospitals, Morgantown, West Virginia
  - Community Comprehensive Cancer Center at Camden-Clark Memorial Hospital, Parkersburg, West Virginia
  - Marshfield Clinic - Chippewa Center, Chippewa Falls, Wisconsin
  - Marshfield Clinic Cancer Care at Regional Cancer Center, Eau Claire, Wisconsin
  - Vince Lombardi Cancer Clinic - Green Bay at Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Gundersen Lutheran Center for Cancer and Blood, La Crosse, Wisconsin
  - Marshfield Clinic - Marshfield Center, Marshfield, Wisconsin
  - Saint Joseph's Hospital, Marshfield, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
  - Medical College of Wisconsin Cancer Center, Milwaukee, Wisconsin
  - Marshfield Clinic - Lakeland Center, Minocqua, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - Ministry Medical Group at Saint Mary's Hospital, Rhinelander, Wisconsin
  - Marshfield Clinic - Indianhead Center, Rice Lake, Wisconsin
  - Marshfield Clinic at Saint Michael's Hospital, Stevens Point, Wisconsin
  - Marshfield Clinic - Wausau Center, Wausau, Wisconsin
  - Aurora Women's Pavilion of West Allis Memorial Hospital, West Allis, Wisconsin
  - Marshfield Clinic - Weston Center, Weston, Wisconsin
  - Marshfield Clinic - Wisconsin Rapids Center, Wisconsin Rapids, Wisconsin
  - Welch Cancer Center at Sheridan Memorial Hospital, Sheridan, Wyoming
- Canada (9):
  - Edmond Odette Cancer Centre at Sunnybrook, Toronto, Ontario
  - Hopital Notre-Dame du CHUM, Montreal, Quebec
  - CHUM - Hotel Dieu Hospital, Montreal, Quebec
  - CHUM - Hopital Saint-Luc, Montreal, Quebec
  - Royal Victoria Hospital - Montreal, Montreal, Quebec
  - Montreal General Hospital, Montreal, Quebec
  - Jewish General Hospital - Montreal, Montreal, Quebec
  - St. Mary's Hospital Center, Montreal, Quebec
  - Hopital du Saint-Sacrement - Quebec, Québec, Quebec
- San Juan City Hospital, San Juan, Puerto Rico

REFERENCES:
- [Result] Bear HD, Tang G, Rastogi P, Geyer CE Jr, Robidoux A, Atkins JN, Baez-Diaz L, Brufsky AM, Mehta RS, Fehrenbacher L, Young JA, Senecal FM, Gaur R, Margolese RG, Adams PT, Gross HM, Costantino JP, Swain SM, Mamounas EP, Wolmark N. Bevacizumab added to neoadjuvant chemotherapy for breast cancer. N Engl J Med. 2012 Jan 26;366(4):310-20. doi: 10.1056/NEJMoa1111097. PMID 22276821
- [Result] Bear HD, Tang G, Rastogi P, et al.: The effect on pCR of bevacizumab and/or antimetabolites added to standard neoadjuvant chemotherapy: NSABP protocol B-40. [Abstract] J Clin Oncol 29 (Suppl 15): A-LBA1005, 2011.
- [Derived] Bear HD, Tang G, Rastogi P, Geyer CE Jr, Liu Q, Robidoux A, Baez-Diaz L, Brufsky AM, Mehta RS, Fehrenbacher L, Young JA, Senecal FM, Gaur R, Margolese RG, Adams PT, Gross HM, Costantino JP, Paik S, Swain SM, Mamounas EP, Wolmark N. Neoadjuvant plus adjuvant bevacizumab in early breast cancer (NSABP B-40 [NRG Oncology]): secondary outcomes of a phase 3, randomised controlled trial. Lancet Oncol. 2015 Sep;16(9):1037-1048. doi: 10.1016/S1470-2045(15)00041-8. Epub 2015 Aug 10. PMID 26272770

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm 1A: Docetaxel Then AC | Arm 1B Docetaxel + Bev Then AC + Bev | Arm 2A: Docetaxel + Capecitabine Then AC | Arm 2B: Docetaxel + Cape + Bev Then AC + Bev | Arm 3A: Docetaxel + Gem Then AC | Arm 3B: Docetaxel + Gem + Bev Then AC + Bev
Started | 201 | 199 | 204 | 201 | 197 | 204
Completed | 199 | 196 | 204 | 194 | 192 | 201
Not Completed | 2 | 3 | 0 | 7 | 5 | 3
Not completed — No follow up data | 2 | 3 | 0 | 7 | 5 | 3

BASELINE CHARACTERISTICS:
Groups:
- Docetaxel Then AC: Docetaxel then AC
- Docetaxel + Bev Then AC + Bev: Docetaxel + Bev then AC + Bev
- Docetaxel + Capecitabine Then AC: Docetaxel + Capecitabine then AC
- Docetaxel + Cape + Bev Then AC + Bev: Docetaxel + Cape + Bev then AC + Bev
- Docetaxel + Gem Then AC: Docetaxel + Gem then AC
- Docetaxel + Gem + Bev Then AC + Bev: Docetaxel + Gem + Bev then AC + Bev
- Total: Total of all reporting groups
Arm/Group | Docetaxel Then AC | Docetaxel + Bev Then AC + Bev | Docetaxel + Capecitabine Then AC | Docetaxel + Cape + Bev Then AC + Bev | Docetaxel + Gem Then AC | Docetaxel + Gem + Bev Then AC + Bev | Total
Number analyzed (Participants) | 201 | 199 | 204 | 201 | 197 | 204 | 1206
Age, Continuous [Mean (Standard Deviation); unit: years] | 48 (9.1) | 49 (9.6) | 49 (9.8) | 49 (10.4) | 48 (9.9) | 48 (9.8) | 48 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 201 | 199 | 204 | 201 | 197 | 204 | 1206
  Male | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Pathologic Complete Response (pCR) of the Primary Tumor in the Breast
Description: Percentage of patients absent of histologic evidence of invasive tumor cells in the surgical breast specimen.
Time Frame: Time of surgery, on average 6 or 13 months
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Arm 1A: Docetaxel Then AC | Arm 1B Docetaxel + Bev Then AC + Bev | Arm 2A: Docetaxel + Capecitabine Then AC | Arm 2B: Docetaxel + Cape + Bev Then AC + Bev | Arm 3A: Docetaxel + Gem Then AC | Arm 3B: Docetaxel + Gem + Bev Then AC + Bev
Number analyzed (Participants) | 199 | 196 | 204 | 194 | 192 | 201
percentage of patients | 33.7 [27.1 to 40.2] | 31.6 [25.1 to 38.1] | 23.5 [17.7 to 29.4] | 36.1 [29.3 to 42.8] | 27.6 [21.3 to 33.9] | 35.8 [29.2 to 42.4]

2. Secondary Outcome: pCR in the Breast and Nodes
Description: Percentage of patients absent of histologic evidence of invasive tumor cells in the surgical breast specimen and axillary lymph nodes.
Time Frame: Time of surgery, on average 6 or 13 months
Population: Arm 1A there is no follow up data for 3 patients; Arm 1B no follow up date for 6 patients; Arm 2A no follow up data for 1 patient; Arm 2B no follow up data for 11 patients; Arm 3A no follow up data for 9 patients; and Arm 3B no follow up data for 6 patients
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Arm 1A: Docetaxel Then AC | Arm 1B Docetaxel + Bev Then AC + Bev | Arm 2A: Docetaxel + Capecitabine Then AC | Arm 2B: Docetaxel + Cape + Bev Then AC + Bev | Arm 3A: Docetaxel + Gem Then AC | Arm 3B: Docetaxel + Gem + Bev Then AC + Bev
Number analyzed (Participants) | 198 | 193 | 203 | 190 | 188 | 198
percentage of patients | 27.3 [21.3 to 33.6] | 24.4 [18.6 to 30.6] | 18.7 [13.7 to 24.4] | 27.4 [21.2 to 33.8] | 22.9 [17.2 to 29.1] | 30.3 [24.1 to 36.8]

3. Secondary Outcome: Clinical Overall Response (cOR) Following Docetaxel Alone, Docetaxel/Capecitabine, and Docetaxel/Gemcitabine Hydrochloride, With or Without Bevacizumab, as Assessed by Physical Exam at the Completion of the Docetaxel-based Portion of Chemotherapy
Description: Percentages of patients assessed as Clinical Complete Response or Clinical Partial Response according to RECIST.
Time Frame: Assessed at cycle 5 of chemotherapy, on average at 15 weeks
Population: For Arm 1A there is no follow up data for 1 patient; Arm 1B no follow up data for 5 patients; Arm 2A no follow up data for 6 patients; Arm 2B no follow up data for 7 patients; Arm 3A no follow up data for 7 patients; Arm 3B no follow up data for 4 patients
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Arm 1A: Docetaxel Then AC | Arm 1B Docetaxel + Bev Then AC + Bev | Arm 2A: Docetaxel + Capecitabine Then AC | Arm 2B: Docetaxel + Cape + Bev Then AC + Bev | Arm 3A: Docetaxel + Gem Then AC | Arm 3B: Docetaxel + Gem + Bev Then AC + Bev
Number analyzed (Participants) | 200 | 194 | 198 | 194 | 190 | 200
percentage of patients | 77 [70.5 to 82.2] | 87.6 [82.1 to 91.5] | 73.7 [67 to 79.3] | 84 [78.1 to 88.5] | 82.6 [76.5 to 87.3] | 88 [82.6 to 91.8]

4. Secondary Outcome: Clinical Overall Response: cOR as Assessed by Physical Exam at the Completion of the Sequential Chemotherapy Regimens
Description: The percentage of patients assessed by physical exam as Clinical Complete Response or Clinical Partial Response according to RECIST.
Time Frame: Three to four weeks after the last chemotherapy dose on average 6 or 13 months
Population: For Arm 1A there is no follow up data for 2 patients; Arm 1B no follow up data for 4 patients; Arm 2A no follow up data for 5 patients; Arm 2B no follow up data for 8 patients; Arm 3A no follow up data for 5 patients; Arm 3B no follow up data for 4 patients
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Arm 1A: Docetaxel Then AC | Arm 1B Docetaxel + Bev Then AC + Bev | Arm 2A: Docetaxel + Capecitabine Then AC | Arm 2B: Docetaxel + Cape + Bev Then AC + Bev | Arm 3A: Docetaxel + Gem Then AC | Arm 3B: Docetaxel + Gem + Bev Then AC + Bev
Number analyzed (Participants) | 199 | 195 | 199 | 193 | 192 | 200
percentage of patients | 79.9 [73.6 to 84.8] | 87.7 [82.2 to 91.6] | 75.4 [68.8 to 80.8] | 90.7 [85.6 to 94] | 83.3 [77.3 to 87.9] | 80.5 [74.3 to 85.4]

5. Secondary Outcome: Clinical Complete Response (cCR) Following Docetaxel Alone, Docetaxel/Capecitabine, and Docetaxel/Gemcitabine Hydrochloride, With or Without Bevacizumab, as Assessed by Physical Exam at Completion of Therapy
Description: Percentages of patients assessed as Clinical Complete Response or Clinical Partial Response according to RECIST.
Time Frame: Assessed at cycle 5 of chemotherapy, on average at 15 weeks
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Arm 1A: Docetaxel Then AC | Arm 1B Docetaxel + Bev Then AC + Bev | Arm 2A: Docetaxel + Capecitabine Then AC | Arm 2B: Docetaxel + Cape + Bev Then AC + Bev | Arm 3A: Docetaxel + Gem Then AC | Arm 3B: Docetaxel + Gem + Bev Then AC + Bev
Number analyzed (Participants) | 199 | 195 | 199 | 193 | 192 | 200
percentage of patients | 30 [23.8 to 36.4] | 43.3 [36.3 to 50.1] | 29.8 [23.6 to 36.2] | 34.5 [27.9 to 41.2] | 37.9 [31 to 44.7] | 42 [35.1 to 48.7]

6. Secondary Outcome: Clinical Complete Resonse: cCR as Assessed by Physical Exam at the Completion of the Sequential Chemotherapy Regimens
Description: The percentage of patients assessed by physical exam as Clinical Complete Response according to RECIST.
Time Frame: Three to four weeks after the last chemotherapy dose, on average at 6 or 13 months
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Arm 1A: Docetaxel Then AC | Arm 1B Docetaxel + Bev Then AC + Bev | Arm 2A: Docetaxel + Capecitabine Then AC | Arm 2B: Docetaxel + Cape + Bev Then AC + Bev | Arm 3A: Docetaxel + Gem Then AC | Arm 3B: Docetaxel + Gem + Bev Then AC + Bev
Number analyzed (Participants) | 199 | 195 | 199 | 193 | 192 | 200
percentage of patients | 52.3 [45.1 to 58.9] | 64.6 [57.5 to 70.9] | 51.3 [44.1 to 57.9] | 59.1 [51.8 to 65.6] | 52.6 [45.3 to 59.4] | 60 [52.9 to 66.4]

7. Secondary Outcome: Percentage of Cardiac Events
Time Frame: After each cycle, 3-5 weeks postoperative, 9 and 12 months from study entry, every 6 month years 2-5, and annually years 6-10, for postoperative bevacizumab patients, every 6 weeks during postoperative therapy and at 18 months following study entry.
Reporting Status: Not Posted

8. Secondary Outcome: Surgical Complication
Description: Number of patients with Grade 4 or above surgery-related toxicities
Time Frame: 24 months after study entry
Population: For Arm 1A there is no follow up data for 8 patients; Arm 1B no follow up data for 8 patients; Arm 2A no follow up data for 6 patients; Arm 2B no follow up data for 12 patients; Arm 3A no follow up data for 11 patients; Arm 3B no follow up data for 7 patients
Measure: Number; unit: participants
Arm/Group | Arm 1A: Docetaxel Then AC | Arm 1B Docetaxel + Bev Then AC + Bev | Arm 2A: Docetaxel + Capecitabine Then AC | Arm 2B: Docetaxel + Cape + Bev Then AC + Bev | Arm 3A: Docetaxel + Gem Then AC | Arm 3B: Docetaxel + Gem + Bev Then AC + Bev
Number analyzed (Participants) | 193 | 191 | 198 | 189 | 186 | 197
participants | 1 | 1 | 0 | 1 | 0 | 1

9. Secondary Outcome: Toxicities Including Events Other Than Congestive Heart Failure, of Chemotherapy Alone, Bevacizumab With Chemotherapy, and Bevacizumab Alone
Description: The number of patients who experienced Grade 1 or above Adverse Events. Referring to the Adverse Events tables for specifics.
Time Frame: 24 months after study entry
Population: For Arm 1A there is no followup data for 2 patients; for Arm 2A there is no followup data for 1 patient; for Arm 3A there is no followup data for 3 patients; for Arm 1B there is no followup data for 3 patients; for Arm 2B there is no followup data for 5 patients; and for Arm 3B there is no followup data for 2 patients.
Measure: Number; unit: participants
Arm/Group | Arm 1A: Docetaxel Then AC | Arm 1B Docetaxel + Bev Then AC + Bev | Arm 2A: Docetaxel + Capecitabine Then AC | Arm 2B: Docetaxel + Cape + Bev Then AC + Bev | Arm 3A: Docetaxel + Gem Then AC | Arm 3B: Docetaxel + Gem + Bev Then AC + Bev
Number analyzed (Participants) | 199 | 196 | 203 | 196 | 194 | 202
participants | 180 | 157 | 172 | 185 | 158 | 185

10. Secondary Outcome: Disease-free Survival (DFS)
Description: Percentage of patients free from local recurrence following mastectomy, local recurrence in the ipsilateral breast following lumpectomy, regional recurrence, distant recurrence, contralateral breast cancer, second primary cancer after 5 years.
Time Frame: Measured through 5 years after study enrollment
Population: For Arm 1A there is no follow up data for 2 patients; Arm 1B no follow up data for 4 patients; Arm 2B no follow up data for 6 patients; Arm 3A no follow up data for 7 patients; Arm 3B no follow up data for 3 patients
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Arm 1A: Docetaxel Then AC | Arm 1B Docetaxel + Bev Then AC + Bev | Arm 2A: Docetaxel + Capecitabine Then AC | Arm 2B: Docetaxel + Cape + Bev Then AC + Bev | Arm 3A: Docetaxel + Gem Then AC | Arm 3B: Docetaxel + Gem + Bev Then AC + Bev
Number analyzed (Participants) | 199 | 195 | 204 | 195 | 190 | 201
percentage of patients | 73.4 [66.2 to 79.3] | 72.2 [65.1 to 78.1] | 68.5 [61 to 74.9] | 77.1 [69.7 to 82.9] | 72.9 [65.3 to 79.1] | 74.8 [66.1 to 81.5]

ADVERSE EVENTS:
Description: Participants at Risk includes any patient who submitted an AE form.
Arm/Group | Docetaxel Then AC | Docetaxel + Bev Then AC + Bev | Docetaxel + Capecitabine Then AC | Docetaxel + Cape + Bev Then AC + Bev | Docetaxel + Gem Then AC | Docetaxel + Gem + Bev Then AC + Bev
Serious Adverse Events (participants affected / at risk) | 4/199 | 15/196 | 8/203 | 30/196 | 2/194 | 15/202
Other Adverse Events (participants affected / at risk) | 118/199 | 150/196 | 168/203 | 182/196 | 150/194 | 178/202
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Docetaxel Then AC (N=199) | Docetaxel + Bev Then AC + Bev (N=196) | Docetaxel + Capecitabine Then AC (N=203) | Docetaxel + Cape + Bev Then AC + Bev (N=196) | Docetaxel + Gem Then AC (N=194) | Docetaxel + Gem + Bev Then AC + Bev (N=202)
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Anaphylaxis (Immune system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Anemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 1
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Cardiac troponin I increased (Investigations) | 0 | 0 | 1 | 1 | 0 | 1
Colonic hemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Colonic perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 2
Depression (Psychiatric disorders) | 0 | 1 | 1 | 1 | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 0 | 1
Endocarditis infective (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0 | 1
Headache (Nervous system disorders) | 0 | 1 | 0 | 1 | 0 | 0
Heart failure (Cardiac disorders) | 0 | 1 | 0 | 1 | 0 | 1
Hyperkalemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0 | 1 | 0 | 0
Hypokalemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 2 | 1 | 1
Hyponatremia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0
Infections and infestations - Other, specify (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Investigations - Other, specify (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 1
Myositis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Nervous system disorders - Other, specify (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 2
Pericardial effusion (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 4 | 0 | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Small intestinal perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 0 | 0
Sudden death NOS (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Thromboembolic event (Vascular disorders) | 1 | 1 | 2 | 4 | 0 | 1
Uterine hemorrhage (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0
Vascular disorders - Other, specify (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 3 | 0 | 2
Leukemia secondary to oncology chemotherapy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0
Treatment related secondary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Visceral arterial ischemia (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0
Anal hemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pleural hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Abdominal infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Lung infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Left ventricular systolic dysfunction (Cardiac disorders) | 0 | 1 | 1 | 5 | 0 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Docetaxel Then AC (N=199) | Docetaxel + Bev Then AC + Bev (N=196) | Docetaxel + Capecitabine Then AC (N=203) | Docetaxel + Cape + Bev Then AC + Bev (N=196) | Docetaxel + Gem Then AC (N=194) | Docetaxel + Gem + Bev Then AC + Bev (N=202)
Alanine aminotransferase increased (ALT/SGPT) (Investigations) | 2 | 9 | 10 | 7 | 26 | 35
Aspartate aminotransferase increased (AST/SGOT) (Investigations) | 3 | 7 | 5 | 8 | 18 | 27
Bone pain (Musculoskeletal and connective tissue disorders) | 10 | 16 | 1 | 7 | 6 | 4
Diarrhea (Gastrointestinal disorders) | 26 | 27 | 52 | 43 | 41 | 43
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 11 | 10 | 5 | 9 | 11 | 14
Fatigue (General disorders) | 18 | 18 | 21 | 21 | 14 | 22
Febrile neutropenia (Blood and lymphatic system disorders) | 5 | 18 | 14 | 23 | 16 | 19
Headache (Nervous system disorders) | 1 | 7 | 2 | 7 | 2 | 11
Hyperglycemia (Metabolism and nutrition disorders) | 11 | 3 | 6 | 3 | 5 | 5
Hypertension (Vascular disorders) | 4 | 49 | 3 | 43 | 2 | 49
Infections and infestations - Other, specify (Infections and infestations) | 4 | 11 | 8 | 16 | 7 | 20
Mucositis oral (Gastrointestinal disorders) | 22 | 54 | 56 | 83 | 38 | 58
Myalgia (Musculoskeletal and connective tissue disorders) | 10 | 9 | 3 | 11 | 4 | 3
Nausea (Gastrointestinal disorders) | 4 | 9 | 8 | 10 | 13 | 9
Neutrophil count decreased (Investigations) | 28 | 30 | 42 | 37 | 64 | 70
Peripheral motor neuropathy (Nervous system disorders) | 8 | 4 | 3 | 13 | 4 | 4
Peripheral sensory neuropathy (Nervous system disorders) | 33 | 35 | 29 | 40 | 19 | 21
Proteinuria (Renal and urinary disorders) | 0 | 12 | 0 | 5 | 0 | 10
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 22 | 22 | 11 | 29 | 33 | 38
Vomiting (Gastrointestinal disorders) | 6 | 4 | 9 | 7 | 16 | 8
White blood cell decreased (Investigations) | 6 | 14 | 14 | 7 | 22 | 16
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 13 | 32 | 92 | 110 | 5 | 14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less